CLINICAL TRIAL: NCT04411706
Title: a Phase II, Open-label, Single Arm Study of Sintilimab (an Anti-PD-1 Inhibitor) Combined With Apatinib and Capecitabine in Advanced Hepatocellular Carcinoma
Brief Title: A Study of Sintilimab Combined With Apatinib and Capecitabine in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTGU005
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Apatinib+Capecitabine (Experimental): =Drug: Sintilimab（i.v）+apatinib（p.o）+capecitabine（p.o）
  Interventions: Drug: Sintilimab Combined With Apatinib and Capecitabine

INTERVENTIONS:
Drug: Sintilimab Combined With Apatinib and Capecitabine — Drug: Sintilimab 200mg (3mg/kg for underweight patients) intravenously, every 21 days for a cycle;
  Drug: Apatinib,250mg po qd, for continuous medication;
  Drug: Capecitabine,1000mg/m2 po bid, d1-d14, every 21 days for a cycle;

SUMMARY:
This study aims to evaluate the efficacy and safety of Sintilimab (an Anti-PD-1 Inhibitor) combined with apatinib and capecitabine as first-line therapy in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given written informed consent.
2. Age between 18-75 years old.male or female.
3. Conform to the clinical diagnosis standard strictly or histological or cytological confirmation of HCC(hepatocellular carcinoma) and with at least one measurable lesion by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to RECIST 1.1 standard.
4. Subjects haven't received any systemic treatment that includes target-therapy, immunotherapy or chemotherapy for HCC before admission.
5. liver function status Child-Pugh Class A; Barcelona Clinic Liver Cancer(BCLC) staging is stage B or C；
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1；
7. Expected survival ≥12 weeks
8. The main organ's function is normal and it should meet the following criteria(Excludes use of any blood components and cell growth factors during the screening period):

   1. Absolute neutrophil count≥1.5×109 /L
   2. Platelets≥80×109/L ;Hemoglobin≥9.0 g/dL; Serum albumin≥3g/dL
   3. Total bilirubin (TBIL)≤1.5×upper limit of normal (ULN); ALT and AST≤1.5×upper limit of normal(ULN); AKP≤ 2.5×upper limit of normal(ULN)
   4. Thyroid stimulating hormone (TSH)≤1.0×upper limit of normal(ULN)（If abnormal, T3 and T4 levels should be examined at the same time）
   5. Serum creatinine ≤1.5×ULN or creatinine clearance > 50 mL/minute (using Cockcroft-Gault formula)

Exclusion Criteria:

1. Patients must not have had prior treatment with Sintilimab or any other PD-L1 or PD-1 antagonists.
2. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
3. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration. Note: corticosteroids used for the purpose of IV contrast allergy prophylaxis are allowed.
4. Known history of hypersensitivity to any components of the Sintilimab formulation, or other antibody formulation.
5. Active central nervous system (CNS) metastases with clinical symptoms (including cerebral edema, steroid requirement, or progressive disease).
6. Patients with other malignant tumor (except cured skin basal cell carcinoma and cervical carcinoma).
7. Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention, left ventricular ejection fraction(LVEF) < 50%.
8. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents(within 3 months): systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg.
9. Coagulation abnormalities (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or are receiving thrombolytic or anticoagulant therapy. Patients with or previous with serious hemorrhage (bleeding > 30 ml within 3 months), haemoptysis (> 5 ml within 4 weeks) of thromboembolic events within 12 months (including stroke events and/or transient ischemic attack).
10. Previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency, such as: esophageal varices, local active ulcerative lesions, gastric ulcer and duodenal ulcer, the ulcerous colitis, gastrointestinal diseases such as portal hypertension or resection of tumor with bleeding risk, etc.
11. Objective evidence of previous or current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, pulmonary function damaged seriously etc.
12. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or active hepatitis (transaminase does not meet the inclusion, hepatitis B virus (HBV) DNA ≥10⁴ /ml or hepatitis C virus (HCV) RNA≥103 /ml or higher)
13. Participated in other clinical trials, or finish other clinical trials within 4 weeks. Patients who may receive other anti-tumor systemic chemotherapy during the study.
14. Patients who may receive vaccination during the study, or previous had vaccination within 4 weeks.
15. Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-06-21 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 year after the last patient's enrollment
  Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 1 year after the last patient's enrollment
  Disease Control Rate (DCR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Duration of Response (DoR) | 1 year after the last patient's enrollment
  Duration of Response (DoR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Overall survival(OS) | 1 year after the last patient's enrollment
  the date of Death of any causes since the date of enrollment
Progression-free survival(PFS) | 1 year after the last patient's enrollment
  Progression-free survival(PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Safety as measured by the rate of AEs | 1 year after the last patient's enrollment
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, Hubei, China

REFERENCES:
- [Derived] Li D, Xu L, Ji J, Bao D, Hu J, Qian Y, Zhou Y, Chen Z, Li D, Li X, Zhang X, Wang H, Yi C, Shi M, Pang Y, Liu S, Xu X. Sintilimab combined with apatinib plus capecitabine in the treatment of unresectable hepatocellular carcinoma: A prospective, open-label, single-arm, phase II clinical study. Front Immunol. 2022 Aug 26;13:944062. doi: 10.3389/fimmu.2022.944062. eCollection 2022. PMID 36091003